CLINICAL TRIAL: NCT06041750
Title: Predicting Postoperative Pulmonary Complications In Obstructive Sleep Apnea Patients; Multicentre, Prospective, Observational Cohort Study
Brief Title: Postoperative Pulmonary Complications In Obstructive Sleep Apnea Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Acibadem University (Other); Baskent University (Other); Celal Bayar University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Assistant Professor, Cukurova University
Other Study IDs: POPCSA
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Obstructive Sleep Apnea; Postoperative Complications
Keywords: obstructive sleep apnea; postoperative pulmonary complications; general anesthesia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSAS patients with postoperative pulmonary complication: American Society of Anesthesiologists (ASA) physical status I-III adult patients age between 18-65 years undergoing elective surgery with general anesthesia and diagnosis of OSAS will be recruited in this study. In this patient group, the incidence of postoperative early-period and long-term pulmonary complications will be investigated.
  Interventions: Procedure: Elective surgical procedure under general anesthesia

INTERVENTIONS:
Procedure: Elective surgical procedure under general anesthesia — The incidence of postoperative pulmonary complications in OSAS patients undergoing elective surgery under general anesthesia will be determined.

SUMMARY:
It is known that perioperative respiratory complications occur more often in obstructive sleep apnea syndrome (OSAS) patients during general anesthesia. Although there are prospective RCTs in this area, the need for further and larger studies remains due to the heterogenity of the results. Moreover, the incidence of postoperative pulmonary complications in OSAS patients undergoing surgery in Turkey and the predictive factors affecting the respiratory adverse events are uncertain. Therefore, in this prospective observational cohort study, it was aimed to determine the incidence of postoperative pulmonary complications and the predictor factors associated with patient, anesthesia and surgery in surgical patients with a confirmed or highly suspected OSAS diagnosis undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years
2. ASA physical status I-III
3. Preoperative OSAS diagnosis (with polysomnography or STOP-BANG questionnaire score)
4. Surgeries performed under general anesthesia
5. Endotracheal intubation facilitated by neuromuscular blockers

Exclusion Criteria:

1. ASA physical status IV or V
2. Planned admission to the ICU after surgery
3. Cardiac Surgery
4. Non-operating room anesthesia
5. Neuromuscular disease
6. Emergency or re-operational procedure
7. Laryngectomy
8. Pneumonectomy
9. Invasive airway access
10. Pregnancy
11. Outpatient surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA status I-III adult patients age between 18-65 years undergoing elective surgery with general anesthesia and diagnosis of OSAS will be recruited in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | Postoperative day 1, 2, 7 and 30.
  The rate of postoperative hypoxia (respiratory failure), atelectasis, pulmonary edema /embolus, aspiration, bronchospasm, respiratory infection / pneumonia, pleural effusion, pneumothorax, respiratory arrest will be measured

SECONDARY OUTCOMES:
Predictive factors | Postoperative day 1, 2, 7 and 30.
  Determination of patient, anesthesia and surgery-related predictive factors affecting the development of postoperative pulmonary complications.
Non-invasive/invasive mechanical ventilation requirement | Postoperative day 1, 2, 7 and 30.
  Determination of the need for non-invasive or invasive mechanical ventilation beyond clinical standards.
Intensive care unit admission | Postoperative day 1, 2, 7 and 30.
  Intensive care unit admission for respiratory indication
Mortality | Postoperative day 30.
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Tütüncü, Prof. Dr., Study Director — İstanbul University, Cerrahpaşa, Faculty of Medicine; Demet Laflı Tunay, Dr., Principal Investigator — Çukurova University, Faculty of Medicine
Locations (1):
- Cukurova University, Adana, Sariçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized by the local researcher. Therefore, data collection will be pseudonymous and the patient's name will not appear on any case report form or other study document. All collected data will be kept confidential. This study will be conducted in accordance with the revision of the Declaration of Helsinki (2008). ICH-GCP will be strictly adhered to.